CLINICAL TRIAL: NCT05976295
Title: Efficacy of Jianpi Qushi Huatan Decoction in the Treatment of Polycystic Ovary Syndrome: A Randomized Double-blind Placebo-controlled Trial
Brief Title: Efficacy of Jianpi Qushi Huatan Decoction in the Treatment of Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ruining Liang, Chief physician, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20223BBG71012-2
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy group (Experimental)
  Interventions: Drug: Jianpi Qushi Huatan Decoction
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jianpi Qushi Huatan Decoction — The treatment group will receive the Jianpi Qushi Huatan Decoction (consisting of Radix astragali, Atractylodes Lancea, Dioscorea oppositifolia, Cyperus rotundus, Lindera aggregata, Aconitum gymnandrum and Ligusticum wallichii, among others). Subjects will take the medication from the first day of inclusion, dissolving and consuming one packet twice a day (morning and evening) for a total of three months.
  Arms: Therapy group
Drug: Placebo — The control group will receive a placebo treatment.
  Arms: Control group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common reproductive disease associated with endocrine and metabolic disorders. Some studies have shown that Chinese herbal medicine is beneficial for PCOS, but the efficacy of Chinese herbal medicine in the treatment of PCOS is not clear, because the quantity of pre-clinical data was limited and the quality of clinical evidence was variable. Therefore, this randomized double-blind placebo-controlled trial aim to evaluate the efficacy of Chinese herbal medicine (Jianpi Qushi Huatan Decoction) in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of PCOS is based on the Rotterdam criteria.
2. Meet the syndrome differentiation standard of spleen deficiency and phlegm-dampness in TCM theory.
3. women aged 18-40 years without fertility requirements.
4. A willingness to undergo this treatment plan.

Exclusion Criteria:

1. Hyperprolactinemia (2 times serum prolactin levels of more than 25 ng/ml at least one week apart).
2. Diminished ovarian reserve, FSH (follicle-stimulating hormone) level more than 10 IU/L.
3. Abnormal thyroid function, TSH (thyroid stimulating hormone) level less than 0.2 mIU/mL or more than 5.5 mIU/mL.
4. Suspected Cushing's syndrome.
5. Adrenal or ovarian tumors secreting androgen.
6. Poorly controlled type II diabetes.
7. Pregnancy or lactation.
8. Hypertensive patients with poorly controlled blood pressure (a systolic blood pressure more than 160 mmHg or a diastolic blood pressure more than 100 mmHg).
9. Those who had taken hormones or other drugs during the previous 3 months.
10. Acute heart, liver, kidney or blood diseases.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Ovulation rate | 3 months
  Ovulation rate in each group during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China